CLINICAL TRIAL: NCT06755125
Title: Effects of KinesioTaping Versus Dry Needling in the Treatment of Sacroiliac Joint Pain Among Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-UOL-SMC/001-31/2024
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Sacroiliac Joint Pain
Keywords: sacroiliac joint pain; piriformis muscle syndrome; acupunture
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping treatment group (Experimental): Patients in Group A were treated with a hot pack, TENS, simple piriformis stretching, and isometric exercises, along with kinesio taping. Kinesio tape was applied directly to the muscle with 50% stretch. During the treatment, kinesio tape was applied to the patients twice a week, for a total of eight applications.
  Interventions: Other: Kinesio Taping
- Dry Needling treatment group (Experimental): Patients in Group B was treated with a hot pack, TENS, simple piriformis stretch, and isometrics, along with Dry Needling of piriformis muscle. During the treatment, Dry Needling was applied to the patients twice a week, eight times in total.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Kinesio Taping — Patients in Group A was treated with a hot pack, TENS, simple piriformis stretch, and isometrics, along with kinesio taping. Kinesio tape was applied directly to the muscle with 50% stretching.During the treatment, kinesio tape will be applied to the patients twice a week, eight times in total.
  Arms: Kinesio taping treatment group
Other: Dry Needling — Patients in Group B was treated with a hot pack, TENS, simple piriformis stretch, and isometrics, along with dry needling.During the treatment, dry needling was applied to the patients twice a week, eight times in total.
  Arms: Dry Needling treatment group

SUMMARY:
The goal of this randomized controlled trial was to investigate the effects of kinesio taping and dry needling on sacroiliac joint (SIJ) pain due to piriformis muscle tightness among females aged 20 to 50 years.

The main research questions it aimed to answer were:

Null Hypothesis (H₀):

There was no significant difference in the effectiveness of kinesio taping and dry needling on SIJ pain caused by piriformis muscle tightness.

Alternate Hypothesis (H₁):

There was a significant difference in the effectiveness of kinesio taping and dry needling on SIJ pain caused by piriformis muscle tightness.

All study participants provided both written and verbal consent. The research was prospective and randomized. The investigation was conducted on individuals between the ages of 20 and 50 during follow-up visits. According to the inclusion and exclusion criteria, a total of 45 participants were selected. Subjects who agreed to participate were randomly assigned to two groups.

Group A received a hot pack, TENS, piriformis simple stretching and isometric exercises, along with kinesio taping.

Group B received a hot pack, TENS, simple stretching and isometric exercises, along with dry needling.

Piriformis tightness was diagnosed using the Piriformis test, and by assessing hip internal rotation and adduction. Sacroiliac joint pain was detected using the Posterior Pain Provocation Test, Gaenslen's Test, and Patrick's Test. At the beginning of the treatment, all participants underwent pretest measurements using the Numeric Pain Rating Scale, Goniometer, Functional Gait Assessment, and Oswestry Disability Index.

DETAILED DESCRIPTION:
All research participants were fully informed about the goals, duration, treatment protocols used within the boundaries of the study, any potential side effects, and concerns that could arise. All study participants provided both written and verbal consent. The research was prospective and randomized. The investigation was conducted on individuals between the ages of 20 and 50 during follow-up visits. According to the inclusion and exclusion criteria, a total of 45 participants were selected. Subjects who intended to participate were randomly assigned to two groups.

Group A received hot packs, TENS, piriformis simple stretching and isometrics, along with the use of kinesio taping.

Group B received hot packs, TENS, simple stretching and isometrics, along with the use of dry needling.

Piriformis tightness was diagnosed using the Piriformis test, and by assessing hip internal rotation and adduction, whereas sacroiliac joint pain was detected using the Posterior Pain Provocation Test, Gaenslen's Test, and Patrick's Test. At the beginning of the treatment, all participants underwent pretest measurements using the Numeric Pain Rating Scale, Goniometer, Functional Gait Assessment, and Oswestry Disability Index.

ELIGIBILITY:
Inclusion Criteria:

* Only females were selected for the study.
* NPRS Score was between 5 to 10.
* Patients who were not have undergone surgery for SIJD.
* Patients with pain in the lower back, gluteal and groin area, and lower extremity lasting for more than 4 weeks but less than 1 year were selected.
* Patients with pain in the lower back, gluteal and groin areas, and lower extremities lasting for more than 4 weeks but less than 1 year were selected.

Exclusion Criteria:

* Musculoskeletal and neurological conditions; lumbar canal stenosis,lumbar spine surgery,vertebral fracture,neurological conditions.
* Inflammatory, autoimmune, and gynecological conditions, Active pelvic inflammatory disease,rheumatological diseases,endometriosis.
* Systemic conditions; Cancer,diabetes mellitus,intermittent vascular claudication,skin allergies.
* Phobia of needles.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS): | 2 Weeks
  The NPRS was used to quantify pain intensity through an 11-point numeric continuum. Individuals are prompted to assess their pain levels within a range from 0 (indicating an absence of pain) to 10 (representing the most extreme imaginable pain)
Goniometer: | 2 weeks
  The UG which has a transparent plastic 360° face, two movable arms, and a 1° gradation was used.
Functional Gait Assessment (FGA) | 2 weeks
  The instrument consists of 10-items: gait level surface, changes in gait speed, gait with horizontal head turns, gait with vertical head turns, gait and pivot turn, step over obstacles, gait with narrow base of support, gait with eyes closed, ambulating backwards, and steps. Each item was demonstrated to the participants by one of the raters to facilitate understanding and will graded on a four-point ordinal scale ranging from 0 (severe impairment), 1 (moderate impairment), 2 (mild impairment), to 3 (normal), with a maximum score of 30 points. The higher the score, the better the participant's postural stability during gait.
Oswestry Disability Index (ODI): | 2 weeks
  The ODI is a questionnaire containing 10 items covering disability caused by low back pain. Each item was assessed on a six-level ordinal scale with '0' describing 'no limitation' and '5' describing 'extreme limitation or an inability to function'. The total score is a percentage calculated by the sum of all answers divided by 50 (the maximum possible number of points) and multiplied by 100 as follows: 'Total score = (∑item scores/50) x 100'.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Baddar Dr., DPT, Principal Investigator — Sehat Medical Complex
Locations (1):
- Sehat Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gartenberg A, Nessim A, Cho W. Sacroiliac joint dysfunction: pathophysiology, diagnosis, and treatment. Eur Spine J. 2021 Oct;30(10):2936-2943. doi: 10.1007/s00586-021-06927-9. Epub 2021 Jul 16. PMID 34272605
- [Background] Kiapour A, Joukar A, Elgafy H, Erbulut DU, Agarwal AK, Goel VK. Biomechanics of the Sacroiliac Joint: Anatomy, Function, Biomechanics, Sexual Dimorphism, and Causes of Pain. Int J Spine Surg. 2020 Feb 10;14(Suppl 1):3-13. doi: 10.14444/6077. eCollection 2020 Feb. PMID 32123652
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32123652/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34272605/